CLINICAL TRIAL: NCT03041805
Title: A Prospective Cohort Register Study for Validation of Caprini Score in Patients Undergoing Varicose Vein Surgery
Brief Title: Caprini Score in Venous Surgery: a Prospective Cohort Study
Acronym: CAPSIVS
Status: Recruiting | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Kirill Lobastov, Associated Professor, Pirogov Russian National Research Medical University
Other Study IDs: CAPSIVS
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Venous Thromboembolism; Varicose Veins
Keywords: venous thromboembolism; deep vein thrombosis; pulmonary embolism; varicose veins; surgery; endovenous laser treatment; radiofrequency ablation; ultrasound-guided foam sclerotherapy; register; anticoagulation
MeSH Terms: conditions — Venous Thromboembolism; Varicose Veins; Venous Thrombosis; Pulmonary Embolism | interventions — Sclerotherapy; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: EVLT — Endovenous laser treatment of great saphenous vein, small saphenous vein, accessorial saphenous vein with different laser wavelength and any bare type
Procedure: RFA — Radiofrequency ablation of great saphenous vein, small saphenous vein, accessorial saphenous vein with ClosureFast technique
Procedure: USFS — Ultrasound guided foam sclerotherapy of great saphenous vein, small saphenous vein, accessorial saphenous vein with polidocanol or tetradecyl sulphate of any concentration
Procedure: HL/stripping — High ligation and stripping of great saphenous vein, small saphenous vein, accessorial saphenous vein
Procedure: Miniphlebectomy — Miniphlebectomy of any varicose veins under local, regional or general anaesthesia
Procedure: Sclerotherapy — Foam or liquid sclerotherapy of any varicose veins with polidocanol or tetradecyl sulphate of any concentration
Device: GCS — Graduated compression stockings may be used after procedure by the decision of the doctor
Drug: LMWH — Low-molecular-weight heparin may be used after procedure by the decision of the doctor

SUMMARY:
The aim of the study is to make a validation of Caprini score in patients undergoing varicose veins surgery, especially endovascular procedures (endovascular laser treatment - EVLT, radiofrequency ablation - RFA, ultrasound-guided foam sclerotherapy - USFS) and to identify patients with elevated risk of postoperative venous thromboembolism (VTE) who will benefit from prophylactic anticoagulation.

DETAILED DESCRIPTION:
A prospective cohort study based on the platform of Ongoing Registry of Treatment of Chronic Venous Diseases (NCT03035747). The study will enrol adult patients undergoing any kind of varicose veins surgery with and without any prophylaxis. The patients should be examined for venous thromboembolic complications during 2-4 weeks after the procedure with mandatory duplex ultrasound.

The study will provide following information:

* the rate of asymptomatic DVT after varicose veins surgery
* the rate of symptomatic VTE after varicose veins surgery
* the rate of thermal-induced thrombosis (EHIT) after endovenous thermal ablation
* the ability of Caprini scores to predict VTE after varicose veins surgery
* identification of patients with high risk of VTE who will benefit from prophylaxis, especially with anticoagulation

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* any kind of varicose vein surgery
* follow up for 4 weeks after the procedure
* examination for VTE at 2-4 weeks after the procedure, including duplex ultrasound

Exclusion Criteria:

- lost for follow-up during 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with varicose veins that undergoing any kind of varicose vein surgery.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
any episode of VTE | 0-4 weeks after procedure
  symptomatic or asymptomatic, confirmed by instrumental diagnostics

SECONDARY OUTCOMES:
symptomatic deep vein thrombosis | 0-4 weeks after procedure
  symptomatic deep vein thrombosis confirmed by duplex ultrasound
symptomatic pulmonary embolism | 0-4 weeks after procedure
  symptomatic pulmonary embolism confirmed by perfusion isotope scanning or CT pulmonary angiography
asymtomatic deep vein thrombosis | 2-4 weeks after procedure
  asymptomatic DVT revealed by duplex ultrasound
endovenous thermal-induced thrombosis | 0-4 weeks after procedure
  EHIT revealed by duplex ultrasound
major bleeding | 0-4 weeks after procedure
  Fatal bleeding, and/or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a fall in haemoglobin level of 20 g/L or more, or leading to transfusion of two or more units of whole blood or red cells.
clinicaly relevant bleeding | 0-4 weeks after procedure
  any non-major bleeding need for treatment or intervention
death for any reason | 0-4 weeks after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kirill Lobastov, PhD, Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No